CLINICAL TRIAL: NCT01513122
Title: Bone and Body Comp: A Sub Study of the SECOND-LINE Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2L body comp sub-study
Record Dates: First submitted 2012-01-16; First posted 2012-01-20 (Estimated); Results first posted 2014-01-17 (Estimated); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: HIV
MeSH Terms: interventions — Lopinavir; Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1. Lopinavir / ritonavir + 2-3N(t)RTI (Active Comparator): LPV/r 200mg/50mg 4 tabs once daily or 2 tabs twice daily + 2-3N(t)RTI
  Interventions: Drug: Lopinavir / ritonavir; Drug: 2-3N(t)RTI
- Arm 2. Lopinavir /ritonavir + raltegravir (Active Comparator)
  Interventions: Drug: Lopinavir / ritonavir; Drug: raltegravir

INTERVENTIONS:
Drug: Lopinavir / ritonavir — LPV/r 200mg/50mg 4 tabs once daily or 2 tabs twice daily
Drug: 2-3N(t)RTI
  Arms: Arm 1. Lopinavir / ritonavir + 2-3N(t)RTI
Drug: raltegravir — raltegravir 400mg 1 tablet twice daily.
  Arms: Arm 2. Lopinavir /ritonavir + raltegravir

SUMMARY:
The use of anti HIV drugs (ART), and in particular a class of drugs known as nucleoside reverse transcriptase inhibitors (N(t)RTI), has been associated with changes in body fat and in particular loss of peripheral fat in the limbs. Low bone mineral density and osteoporosis are also common in HIV-infected patients. There appears to be some association between ART and bone loss, but this is poorly understood and requires further research. The SECOND-LINE study provides an opportunity to examine if a new anti-HIV drug (raltegravir) can result in greater increase in limb fat than a drug regimen containing N(t)RTI, which is currently standard of care. This study also provides an opportunity to examine if additional bone loss occurs with the second regimen of anti-HIV drugs and whether non-N(t)RTI regimens of ART used in second line therapy result in more or less bone loss than use of other classes of anti-HIV drugs such as protease inhibitors or N(t)RTI combinations.

It is hypothesized that subjects randomised into Raltegravir arm will demonstrate greater increases in limb fat and smaller reductions in bone density at the proximal femur over 48 weeks than those randomised into the control arm (LPV/r + 2-3N(t)RTIs).

ELIGIBILITY:
Second-Line main study identifier: NCT00931463

Inclusion Criteria:

1. HIV-1 positive by licensed diagnostic test
2. Aged 16 years or older (or minimum age as determined by local regulations or as legal requirements dictate)
3. Have received first antiretroviral regimen consisting of an NNRTI plus 2N(t)RTIs for ≥ 24 weeks
4. No change in antiretroviral therapy within 12 weeks prior to screening
5. Failed first-line NNRTI + 2N(t)RTI combination therapy according to virological criteria defined by two consecutive (≥7 days apart) HIV RNA results of > 500 copies/mL
6. No prior or current exposure to HIV protease inhibitors and/or HIV integrase inhibitors
7. Able to provide written informed consent

Exclusion Criteria:

1. The following laboratory variables:

   * absolute neutrophil count (ANC) < 500 cells/µL
   * hemoglobin < 7.0 g/dL
   * platelet count < 50,000 cells/µL
   * ALT > 5 x ULN
2. Pregnant or nursing mothers
3. Participants with active viral hepatitis B infection defined by the presence in serum of hepatitis B surface antigen
4. Use of immunomodulators within 30 days prior to screening
5. Use of any prohibited medications (rifampicin, midazolam, triazolam, cisapride, pimozide, amiodarone, dihydroergotamine, ergotamine, ergonovine, methylergonovine, astemizole, terfenadine, vardenafil, and St. John's wort)
6. Intercurrent illness requiring hospitalisation
7. Active opportunistic disease not under adequate control in the opinion of the site Principal Investigator
8. Participants with current alcohol or illicit substance abuse that in the opinion of the site Principal Investigator might adversely affect participation in the study
9. Participants deemed by the site Principal Investigator unlikely to be able to remain in follow-up for the protocol-defined period

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2010-02; Primary Completion 2012-09 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paddy Mallon, Principal Investigator — Mater Misericordiae University Hospital, Dublin; Waldo Belloso, Principal Investigator — Hospital Italiano, Argentina; Samuel Ferret, Principal Investigator — Hopital Saint-Louis, France; Praphan Phanuphak, Principal Investigator — HIV-NAT Program on AIDS - Thai Red Cross, Bangkok; Jennifer Hoy, Principal Investigator — The Alfred
Locations (7):
- CEADI, Buenos Aires, Argentina
- YRGCare Medical Centre, Chennai, India
- University of Malaya Medical Centre, Kuala Lumpur, Malaysia
- South Africa (3):
  - JOSHA Research, Bloemfontein
  - Desmond Tutu HIV Foundation, Cape Town
  - Chris Hani Baragwanath Hospital, Soweto
- HIV-NAT Program on AIDS - Thai Red Cross, Bangkok, Thailand

REFERENCES:
- [Result] Martin A, Moore C, Mallon PW, Hoy J, Emery S, Belloso W, Phanuphak P, Ferret S, Cooper DA, Boyd MA; Second Line study team. Bone mineral density in HIV participants randomized to raltegravir and lopinavir/ritonavir compared with standard second line therapy. AIDS. 2013 Sep 24;27(15):2403-11. doi: 10.1097/01.aids.0000432534.47217.b4. PMID 23921615
- [Result] Martin A, Moore CL, Mallon PW, Hoy JF, Emery S, Belloso WH, Phanuphak P, Ferret S, Cooper DA, Boyd MA; Second-Line Study Team. HIV lipodystrophy in participants randomised to lopinavir/ritonavir (LPV/r) +2-3 nucleoside/nucleotide reverse transcriptase inhibitors (N(t)RTI) or LPV/r + raltegravir as second-line antiretroviral therapy. PLoS One. 2013 Oct 30;8(10):e77138. doi: 10.1371/journal.pone.0077138. eCollection 2013. PMID 24204757
- [Derived] Boyd MA, Amin J, Mallon PW, Kumarasamy N, Lombaard J, Wood R, Chetchotisakd P, Phanuphak P, Mohapi L, Azwa I, Belloso WH, Molina JM, Hoy J, Moore CL, Emery S, Cooper DA; SECOND-LINE Study Group. Body composition and metabolic outcomes after 96 weeks of treatment with ritonavir-boosted lopinavir plus either nucleoside or nucleotide reverse transcriptase inhibitors or raltegravir in patients with HIV with virological failure of a standard first-line antiretroviral therapy regimen: a substudy of the randomised, open-label, non-inferiority SECOND-LINE study. Lancet HIV. 2017 Jan;4(1):e13-e20. doi: 10.1016/S2352-3018(16)30189-8. Epub 2016 Nov 1. PMID 27815068

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1. Lopinavir / Ritonavir + 2-3N(t)RTI: Lopinavir / ritonavir + 2-3N(t)RTI: LPV/r 200mg/50mg 4 tabs once daily or 2 tabs twice daily + 2-3 N(t)RTI
- Arm 2. Lopinavir /Ritonavir + Raltegravir: Lopinavir /ritonavir + raltegravir: LPV/r 200mg/50mg 4 tabs once daily or 2 tabs twice daily + raltegravir 400mg 1 tablet twice daily.
Period: Overall Study
Arm/Group | Arm 1. Lopinavir / Ritonavir + 2-3N(t)RTI | Arm 2. Lopinavir /Ritonavir + Raltegravir
Started | 102 | 108
Completed | 91 | 105
Not Completed | 11 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1. Lopinavir / Ritonavir + 2-3N(t)RTI | Arm 2. Lopinavir /Ritonavir + Raltegravir | Total
Number analyzed (Participants) | 102 | 108 | 210
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 38.6 (7.8) [34.2 to 44.1] | 38.9 (7.7) [32.6 to 44.4] | 38.8 (7.8) [32.9 to 44.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 63 | 110
  Male | 55 | 45 | 100

OUTCOME MEASURES:

1. Primary Outcome: Mean Bone Mineral Density Changes From Baseline to 48 Weeks as Measured by DXA Scan
Time Frame: 48 weeks
Population: 97 participants reached week 48 in 2-3N(t)RTI arm. 107 reached week 48 in the RAL arm (1 death)
Measure: Mean (95% Confidence Interval); unit: percentage change
Arm/Group | Arm 1. Lopinavir / Ritonavir + 2-3N(t)RTI | Arm 2. Lopinavir /Ritonavir + Raltegravir
Number analyzed (Participants) | 97 | 107
percentage change | -5.2 [-6.7 to -3.8] | -2.9 [-4.3 to -1.5]

2. Primary Outcome: Mean Limbs Fat Changes From Baseline to 48 Weeks as Measured by DXA Scan
Time Frame: 48 weeks
Measure: Mean (95% Confidence Interval); unit: percentage change
Arm/Group | Arm 1. Lopinavir / Ritonavir + 2-3N(t)RTI | Arm 2. Lopinavir /Ritonavir + Raltegravir
Number analyzed (Participants) | 94 | 107
percentage change | 15.7 [5.3 to 25.9] | 21.1 [11.1 to 31.1]

3. Secondary Outcome: Mean Total Body Fat Changes From Baseline to 48 Weeks as Measured by DXA Scan
Time Frame: 48 weeks
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Arm 1. Lopinavir / Ritonavir + 2-3N(t)RTI | Arm 2. Lopinavir /Ritonavir + Raltegravir
Number analyzed (Participants) | 94 | 107
kg | 1.4 [0.2 to 2.7] | 2.1 [0.9 to 3.3]

4. Secondary Outcome: Mean Triglycerides Changes From Baseline to 48 Weeks
Time Frame: 48 weeks
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Arm 1. Lopinavir / Ritonavir + 2-3N(t)RTI | Arm 2. Lopinavir /Ritonavir + Raltegravir
Number analyzed (Participants) | 94 | 105
mmol/L | 0.6 [0.3 to 0.9] | 0.8 [0.6 to 1.0]

5. Secondary Outcome: Mean Total Cholesterol Changes From Baseline to 48 Weeks
Time Frame: 48 weeks
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Arm 1. Lopinavir / Ritonavir + 2-3N(t)RTI | Arm 2. Lopinavir /Ritonavir + Raltegravir
Number analyzed (Participants) | 94 | 105
mmol/L | 0.4 [0.1 to 0.6] | 0.6 [0.4 to 0.9]

6. Secondary Outcome: Mean Glucose Changes From Baseline to 48 Weeks
Time Frame: 48 weeks
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Arm 1. Lopinavir / Ritonavir + 2-3N(t)RTI | Arm 2. Lopinavir /Ritonavir + Raltegravir
Number analyzed (Participants) | 94 | 105
mmol/L | -0.04 [-0.2 to 0.2] | -0.1 [-0.4 to 0.1]

ADVERSE EVENTS:
Description: Adverse Events were not planned to be analyzed for the sub-study and that complete adverse event information is included in the main study report (NCT00931463)
Arm/Group | Arm 1. Lopinavir / Ritonavir + 2-3N(t)RTI | Arm 2. Lopinavir /Ritonavir + Raltegravir
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is a Clinical Trial Agreement signed with each PI detailing the publication policy and disclosure of study's information, in summary:

The Institution, its personnel and the Principal Investigator must not Publish or present any aspect of the Study without the prior written approval of the sponsor, except for the purposes of internal training Publications or presentations of results from the Study will follow the agreement's publication/presentation guidelines